CLINICAL TRIAL: NCT03730415
Title: The Effects of Viscoelastic Guided Transfusions During Severe Thermal Injury Burn Excision on Post Transfusion Infections
Brief Title: The Effects of Viscoelastometry Guided Resuscitation During Burn Excision on Post Resuscitation Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Michael Cripps, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 032014-072
Record Dates: First submitted 2016-05-23; First posted 2018-11-05 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viscoelastic (VE) guided transfusion (Experimental): The intervention made in the VE guided transfusion group is that the VE results will be available to the treating physicians to guide transfusions based on VE results during their burn excision.
  Interventions: Procedure: Viscoelastic (VE) Guided Transfusion
- Standard practice transfusion (No Intervention): The standard practice transfusion group will receive the current standard transfusion practice during their burn excision, which is based solely on physician preference using standard lab values.

INTERVENTIONS:
Procedure: Viscoelastic (VE) Guided Transfusion — A viscoelastic analyzer (ROTEM) will be used to guide the transfusion algorithm during the burn wound excision of subjects enrolled into this arm
  Arms: Viscoelastic (VE) guided transfusion

SUMMARY:
This is a randomized controlled trial to compare viscoelastometric (VE) guided transfusion to standard practice transfusion in severe thermal injury burn excision on the utilization of blood products, effects on coagulation and inflammatory mediators, and how these strategies affect post resuscitation infections.

DETAILED DESCRIPTION:
This is an open labeled study as the viscoelastometric (VE) guided transfusion will be based on the visible VE results. Subjects will be randomized to receive either the standard practice transfusion or VE guided transfusion. Blood samples, standard demographic information, and routine laboratory data will be collected on all subjects in the Burn ICU (BICU) enrolled in the study. VE analysis will be performed on ALL subjects immediately prior to the burn excision, and approximately every 40 minutes while the patient is in the operating room (OR) as well as on arrival to the BICU and every 8 hours depending on their need for ongoing transfusion for a maximum of 24 hours. As our intervention, only the VE based transfusion group will have access to the VE analysis at time of transfusion. The VE results will be used at the discretion of the treating physician based on the VE guided transfusion algorithm. Outcomes include the number and timing of blood products transfused from the time of randomization to 24 hours post randomization and the presence of any 30 day post-transfusion infections.

ELIGIBILITY:
Inclusion Criteria:

* Burn patients admitted to Parkland Hospital with total burn surface area (TBSA) greater than 20%

Exclusion Criteria:

* Patients admitted to Parkland Hospital for reasons other than burns or for burns less than or equal to 20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Number of blood products transfused | 24 hours post randomization
  Compare the number of blood products transfused in VE guided transfusion versus standard practice transfusion in burned patients (TBSA >20%) undergoing burn wound excision will be analyzed.

SECONDARY OUTCOMES:
Coagulation factors | excision to 24 hours post excision
  Compare the effects of VE guided transfusion to standard practice transfusion on the coagulation factor in patients undergoing burn wound excision. Changes in individual coagulation factors will be measured. Will measure other related mediators including coagulation Factors V, VIII, and plasminogen activator inhibitor 1 (PAI-1) which have also been implicated in ATC.
Inflammatory Mediators - plasminogen activator inhibitor 1 | excision to 24 hours post excision
  Compare the effects of VE guided transfusion to standard practice transfusion on the inflammatory mediators in patients undergoing burn wound excision. Changes in inflammatory mediators will be measured. Further, analysis into interactions between these factors will be studied.

OTHER OUTCOMES:
Post transfusion infections | 30 days
  Compare the post transfusion infections to the number of blood products transfused for VE guided transfusion and standard practice transfusion in patients undergoing burn wound excision.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Cripps, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] Schaden E, Kimberger O, Kraincuk P, Baron DM, Metnitz PG, Kozek-Langenecker S. Perioperative treatment algorithm for bleeding burn patients reduces allogeneic blood product requirements. Br J Anaesth. 2012 Sep;109(3):376-81. doi: 10.1093/bja/aes186. Epub 2012 Jun 19. PMID 22719014